CLINICAL TRIAL: NCT00255801
Title: Phase II Trial of Doxorubicin HCl Liposome Injection (Doxil®) in Advanced Stage Cutaneous T-Cell Lymphoma Followed by Bexarotene (Targretin®)
Brief Title: Liposomal Doxorubicin Followed By Bexarotene in Treating Patients With Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Tibotec Pharmaceutical Limited (Industry); M.D. Anderson Cancer Center (Other); NYU Langone Health (Other); Hackensack Meridian Health (Other); Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-098; MSKCC-05098
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Bexarotene

ARMS (1):
- Doxil and Targretin® (bexarotene) (Experimental): Patients will be treated with intravenous Doxil® every two weeks for 8 doses (16 weeks). Responses will be assessed. They will then receive Targretin® (bexarotene) orally for at least 16 weeks. Patients who achieve a CR or PR may continue on Targretin® (bexarotene) until relapse.
  Interventions: Drug: Targretin® (bexarotene); Drug: pegylated liposomal doxorubicin hydrochloride

INTERVENTIONS:
Drug: Targretin® (bexarotene)
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin and bexarotene, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bexarotene may also cause cutaneous T-cell lymphoma cells to look more like normal cells, and to grow and spread more slowly. Giving liposomal doxorubicin followed by bexarotene may be an effective treatment for cutaneous T-cell lymphoma.

PURPOSE: This phase II trial is studying how well giving liposomal doxorubicin followed by bexarotene works in treating patients with cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival of patients with stage IB-IV cutaneous T-cell lymphoma treated with doxorubicin HCl liposome followed by bexarotene.

Secondary

* Determine the complete and partial response rate in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive doxorubicin HCl liposome IV over 30-90 minutes once on day 1. Treatment repeats every 2 weeks for 8 courses. Beginning within 4 weeks after the last dose of doxorubicin HCl liposome, patients receive oral bexarotene once daily for at least 16 weeks. Patients who achieve a complete or partial response may continue to receive bexarotene in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell lymphoma

  * Stage IB-IV disease
* Measurable disease
* Newly diagnosed or previously treated disease

  * No demonstrated resistance to prior bexarotene

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* Ejection fraction ≥ 50% by MUGA or 2-D echocardiogram
* No New York Heart Association class II-IV heart disease
* No clinical evidence of congestive heart failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study treatment
* No history of hypersensitivity reactions attributed to doxorubicin HCl liposome or its components
* No active potentially life-threatening infection
* No other acute disease

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics
* Prior doxorubicin allowed provided the cumulative dose is ≤ 300 mg/m^2
* Prior epirubicin hydrochloride allowed provided the cumulative dose is ≤ 540 mg/m^2

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-11; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Straus, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Steven M. Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Patricia L. Myskowski, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Derived] Straus DJ, Duvic M, Horwitz SM, Hymes K, Goy A, Hernandez-Ilizaliturri FJ, Feldman T, Wegner B, Myskowski PL. Final results of phase II trial of doxorubicin HCl liposome injection followed by bexarotene in advanced cutaneous T-cell lymphoma. Ann Oncol. 2014 Jan;25(1):206-10. doi: 10.1093/annonc/mdt480. Epub 2013 Nov 26. PMID 24285015
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxil and Targretin® (Bexarotene)
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Doxil and Targretin® (Bexarotene)
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 56 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Description: CRITERIA FOR THERAPEUTIC RESPONSE/OUTCOME ASSESSMENT
  * CT scans of chest, abdomen and pelvis for TNM stage IV patients who had positive findings prior to treatment.
  * CBC with Sézary cell count and/or flow cytometry in patients with Sézary syndrome.
  * Dermatologic responses will be determined by the Severity-Weighted Assessment Tool (SWAT), a standardized approach to measuring the extent and severity of overall skin disease in patients with CTCL Primary skin tumor assessments were made by the modified Severity-Weighted Assessment Tool (mSWAT) [12, 13]; the Composite Assessment of Index Lesion Severity (CA) [9, 14] was used a secondary scale. Progression was defined as ≥25% increase in mSWAT skin score and ≥50% increase in the sum of the products of the greatest diameters of involved lymph nodes over baseline for patients with involved lymph nodes with stage IV disease
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Doxil and Targretin® (Bexarotene)
Number analyzed (Participants) | 37
months | 5 [0.16 to 26.26]

2. Secondary Outcome: Maximum Therapeutic Response
Description: as for outcome 1
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Doxil and Targretin® (Bexarotene)
Number analyzed (Participants) | 37
Participants
  Clinical Complete Response | 2
  Partial Response | 12
  Stable Disease | 6
  Progressive Disease | 14
  Not Evaluable | 3

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Doxil and Targretin® (Bexarotene)
All-Cause Mortality (participants affected / at risk) | 12/37
Serious Adverse Events (participants affected / at risk) | 15/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxil and Targretin® (Bexarotene) (N=37)
Cardiac Arrhythmia, other (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastritis (incl bile reflux gastritis) (Gastrointestinal disorders) | 1
Inf norm ANC/gr1/2 neut-Cellulitis(skin) (Infections and infestations) | 1
Inf unknown ANC-Blood (Infections and infestations) | 1
Inf unknown ANC-Cellulitis(skin) (Infections and infestations) | 1
Infection, other (Infections and infestations) | 5
Leukocytes (total WBC) (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Pain - Skin (Skin and subcutaneous tissue disorders) | 1
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonitis/pulm infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rigors/chills (General disorders) | 2
Ulceration (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxil and Targretin® (Bexarotene) (N=37)
Hyperglycemia (Metabolism and nutrition disorders) | 11
White blood cells (Investigations) | 9
Cholesterol, high (Investigations) | 7
Triglyceride, high (Metabolism and nutrition disorders) | 7
Fatigue (General disorders) | 4
Neutrophils (Investigations) | 4
Lymphopenia (Investigations) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-09-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT00255801/Prot_SAP_000.pdf